CLINICAL TRIAL: NCT04284111
Title: A Prospective, Multi-center Study of the Effect of Orthokeratology on Myopia Progression in Chinese Children
Brief Title: A Multi-center Study of the Effect of Orthokeratology on Myopia Progression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ019
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with myopia: A total of 1,000 children from 8 hospitals in China is required to undergo ophthalmic examinations and complete questionnaires at baseline and
  1yr after wearing ortho-k lenses.
  Interventions: Device: Orthokeratology lenses

INTERVENTIONS:
Device: Orthokeratology lenses — Orthokeratology lenses

SUMMARY:
This is a prospective study to validate an algorithm for predicting the effect of orthokeratology on myopia progression in children from 8 hospitals in China.

DETAILED DESCRIPTION:
Orthokeratology (ortho-K) is thought to be an effective way to control the progression of Myopia in children, but its effectiveness may vary among different individuals. The investigators therefore conducted a prospective, multi-center study to use an algorithm to predict the progression of myopia among Chinese children wearing Orthokeratology lenses.

ELIGIBILITY:
Inclusion Criteria:

* -6.0D≤SER≤-0.5D
* Astigmatism≤2.0D

Exclusion Criteria:

* Contraindications of wearing Ortho-K.
* Diagnosis of strabismus, amblyopia and other refractive development of the eye or systemic diseases.
* Currently involved in other clinical studies.

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: 1,000 children from 8 hospitals in China plan to wear orthokeratology lenses for myopia control.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
AUROC of the prediction algorithm for identifying fast progressing myopes | 1 year
  Age-specific axial length (AL) changes previously described by Wang et al.(IOVS, 52 (11), 7949-53, 2011) are used as cut-off values to determine whether a child is a fast progressor or not. A child whose AL change falls on or above the cut-off value is considered to be a fast progressor.

SECONDARY OUTCOMES:
Sensitivity and specificity of the prediction algorithm for identifying fast progressing myopes | 1 year
  The investigators will estimate sensitivity and specificity of the predictive algorithm for identifying fast progressing myopes.
Performance of an algorithm for predicting AL | 1 year
  The investigators will use mean absolute error (MAE), R square to evaluate the performance.
Performance of an algorithm for predicting spherical equivalent refractive error | 1 year
  The investigators will use mean absolute error (MAE), R square to evaluate the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Xialin Liu, M.D. Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (8):
- China (8):
  - Hefei Bright Eye Hospital, Hefei, Anhui
  - Zhongshan Ophthalmic Center (Haizhu Branch), Sun Yat-sen University, Guangzhou, Guangdong
  - Wuhan Bright Eye hospital, Wuhan, Hubei
  - Nanchang Bright Eye Hospital, Nanchang, Jiangxi
  - Jinan Bright Eye Hospital, Jinan, Shandong
  - Shanghai Bright Eye Hospital, Shanghai, Shanghai Municipality
  - Chengdu Bright Eye Hospital, Chengdu, Sichuan
  - Kunming Bright Eye hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Ding X, Liu B, Zhang J, He M. Longitudinal changes of axial length and height are associated and concomitant in children. Invest Ophthalmol Vis Sci. 2011 Oct 10;52(11):7949-53. doi: 10.1167/iovs.11-7684. PMID 21896861